CLINICAL TRIAL: NCT02614508
Title: A Phase I Study of Buparlisib (BKM120) and Ofatumumab or Ibrutinib in Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia
Brief Title: Buparlisib and Ofatumumab or Ibrutinib in Treating Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Jonathon Cohen, Principal Investigator, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00071983; NCI-2015-00652 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship2494-13/CBKM120ZUS36T (Other: Emory University/Winship Cancer Institute)
Record Dates: First submitted 2015-11-23; First posted 2015-11-25 (Estimated); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: Recurrent Chronic Lymphocytic Leukemia; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — NVP-BKM120; ibrutinib; ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort A (buparlisib, ofatumumab) (Experimental): Patients receive buparlisib PO QD on days 1-28 and ofatumumab IV on days 1, 8, 15, and 22 during of courses 1-2; and day 1 of courses 4-7. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Buparlisib; Biological: Ofatumumab
- Cohort B (buparlisib, ibrutinib) (Experimental): Patients receive buparlisib as in Cohort A and ibrutinib PO on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Buparlisib; Drug: Ibrutinib

INTERVENTIONS:
Drug: Buparlisib — Given PO
  Other Names: BKM120; PI3K Inhibitor BKM120
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; PCI-32765
  Arms: Cohort B (buparlisib, ibrutinib)
Biological: Ofatumumab — Given IV
  Other Names: Arzerra; GSK1841157; HuMax-CD20; HuMax-CD20, 2F2
  Arms: Cohort A (buparlisib, ofatumumab)

SUMMARY:
This phase I trial studies the side effects and best dose of buparlisib when given together with ofatumumab or ibrutinib in treating patients with chronic lymphocytic leukemia that has returned after a period of improvement or does not respond to treatment. Buparlisib and ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as ofatumumab, may block cancer growth in different ways by targeting certain cells. Giving buparlisib or ibrutinib and ofatumumab together may work better in treating patients with chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and dose limiting toxicities (DLT) of combined ofatumumab and buparlisib in patients with previously treated chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL) who have been exposed to ibrutinib (i.e., ibrutinib pre-treated).

II. To evaluate the safety and dose limiting toxicities (DLT) of combined ibrutinib and buparlisib in patients with previously treated chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL) who have NOT been exposed to ibrutinib (i.e., ibrutinib naïve)

SECONDARY OBJECTIVES:

I. To determine specific toxicities associated with combined buparlisib and ofatumumab.

II. Evaluate for efficacy of buparlisib in combination with ofatumumab in ibrutinib pre-treated patients with CLL/SLL.

III. To determine specific toxicities associated with combined buparlisib and ibrutinib.

IV. To evaluate for efficacy of buparlisib in combination with ibrutinib in ibrutinib naive patients with CLL/SLL.

OUTLINE: This is a dose escalation study of buparlisib. Patients are assigned to 1 of 2 treatment cohorts.

COHORT A (ibrutinib pre-treated): Patients receive buparlisib orally (PO) once daily (QD) on days 1-28 and ofatumumab intravenously (IV) on days 1, 8, 15, and 22 during of courses 1-2; and day 1 of courses 4-7. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

COHORT B (ibrutinib naive): Patients receive buparlisib as in Cohort A and ibrutinib PO on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed B-cell chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL) according to World Health Organization (WHO) criteria with at least one of the following indications for treatment:

  * Progressive disease or marked splenomegaly or hepatomegaly
  * Anemia (hemoglobin [Hgb] < 11 mg/dL) or thrombocytopenia (platelets < 100,000 /mm³)
  * Unexplained weight loss exceeding 10% of body weight over the preceding 6 months
  * Fevers > 100.5° F or night sweats for greater than 2 weeks without evidence of infection
  * Progressive lymphocytosis, with an increase exceeding 50% over a 2 month period or a doubling time of less than 6 months
  * Significant fatigue (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version [v] 4.03 grade 2 or higher)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* At least one prior therapy for CLL/SLL; prior autologous or allogeneic stem cell transplant is allowed; patients may not be on chronic immunosuppressive therapy for graft-versus-host disease (GVHD); patients who are on only oral steroids must be on an oral dose of 10mg or less of prednisone (or equivalent) daily
* Prior therapy with a selective phosphoinositide 3-kinase (PI3K) inhibitor or other B-cell receptor targeting agents is allowed
* Patients who have been previously treated with ibrutinib (or any Bruton's tyrosine kinase [BTK] inhibitor) are eligible for the ibrutinib pre-treated cohort as long as prior ibrutinib or BTK inhibitor therapy was not discontinued due to toxicity/adverse event; there is no minimum dose of ibrutinib; any prior administration will disqualify patients for the ibrutinib-naïve cohort and will require enrollment on the ibrutinib pre-treated cohort
* Serum creatinine ≤ 1.5 x upper limit of normal (ULN) and/or creatinine clearance > 50% lower limit of normal
* Total bilirubin ≤ upper limit of normal (or ≤ 1.5 x upper limit of normal if live metastases are present; or total bilirubin ≤ 3.0 x upper limit of normal with direct bilirubin within normal range in patients with well documented Gilbert's syndrome, which is defined as presence of several episodes of unconjugated hyperbilirubinemia with normal results from complete blood count [CBC] count [including normal reticulocyte count and blood smear], normal liver function test results, and absence of other contributing disease processes at the time of diagnosis)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ upper limit of normal (or < 3.0 x ULN if liver metastases are present)
* Serum lipase ≤ upper limit of normal
* Serum amylase ≤ upper limit of normal
* International normalized ratio (INR) ≤ 1.5
* Fasting glucose ≤ 120 mg/dL
* Absolute neutrophil count ≥ 1000/mm³
* Platelets ≥ 50,000/mm³
* Potassium within normal limits (oral supplementation is allowed)
* Calcium (corrected for albumin) within normal limits (oral supplementation is allowed)
* Hemoglobin A1c (HbA1c) ≤ 8%
* Recovery to ≤ grade 1 toxicities associated with prior therapy
* Negative serum pregnancy test within 72 hours before starting study treatment in women with childbearing potential
* Patient has signed the informed consent (ICF) prior to any screening procedures being performed and is able to comply with protocol requirement
* Patient is able to swallow and retain oral medication
* Patients with diabetes mellitus are eligible if they require oral agents only and have a fasting blood glucose ≤ 120 mg/dL; patients with a history of diabetes mellitus who require daily long-acting or mealtime insulin are not eligible; patients who have previously required treatment for hyperglycemia due to steroids or other medications are eligible as long as they have not required insulin or any other oral agent within 2 months prior to study enrollment

Exclusion Criteria:

* Patient has a known hypersensitivity to any of the excipients of buparlisib
* Patient who has received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug or who have not recovered to grade 1 or better from related side effects of such therapy (except alopecia)
* Patient has not recovered to grade 1 or better (except alopecia) from related side effects of any prior antineoplastic therapy
* Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects
* Patient is currently receiving increasing or chronic treatment (> 5 days) with corticosteroids or another immunosuppressive agent, as chronic administration of corticosteroids (> 5 days) can induce cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4); see also section "concomitant medication"; the following uses of corticosteroids are permitted: single doses; e.g. with standard premedication for infusions; topical applications (e.g., rash), inhaled sprays (e.g., obstructive airways diseases), eye drops or local injections (e.g., intra-articular); patients may take 10mg or less (or equivalent) of oral prednisone daily
* Patient is being treated at start of study treatment with any of the following drugs:

  * Drugs known to be strong inhibitors or inducers of isoenzyme CYP3A4 including herbal medications
  * Drugs with a known risk to induce Torsades de Pointes
  * Note: the patient must have discontinued strong inducers for at least one week and must have discontinued strong inhibitors before the treatment is initiated; switching to a different medication prior to starting study treatment is allowed
* Patient is currently receiving warfarin or other coumarin derived anti-coagulant, for treatment, prophylaxis or otherwise; therapy with heparin, low molecular weight heparin (LMWH), or fondaparinux is allowed
* Patients who have other concurrent severe and/or uncontrolled medical conditions that would, in the investigator's judgment, contraindicate patient participation in the clinical study (eg. active or uncontrolled severe infection, chronic active hepatitis, immuno-compromised, acute or chronic pancreatitis, uncontrolled high blood pressure, interstitial lung disease, etc.)
* Patient has a known history of human immunodeficiency virus (HIV) infection (testing not mandatory)
* Patients has any of the following cardiac abnormalities:

  * Symptomatic congestive heart failure

    * History of documented congestive heart failure (New York Heart Association functional classification III-IV), documented cardiomyopathy
    * Left ventricular ejection fraction < 50% as determined by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO)
  * Myocardial infarction ≤ 6 months prior to enrollment
  * Unstable angina pectoris
  * Serious uncontrolled cardiac arrhythmia
  * Symptomatic pericarditis
  * Corrected QT interval using Fridericia's formula (QTcF) > 480 msec on the screening electrocardiogram (ECG) (using the QTcF formula)
* Currently receiving treatment with medication that has a known risk to prolong the QT interval or inducing Torsades de Pointes, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug
* Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Patient has a score ≥ 12 on the Patient Health Questionnaire (PHQ)-9 questionnaire
* Patient selects a response of "1, 2 or 3" to question number 9 on the PHQ-9 questionnaire regarding potential for suicidal thoughts or ideation (independent of the total score of the PHQ-9)
* Patient has a Generalized Anxiety Disorder (GAD)-7 mood scale score ≥ 15
* Patient has a medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (e.g. risk of doing harm to self or others), or patients with active severe personality disorders (defined according to Diagnostic and Statistical Manual of Mental Disorders [DSM]- IV) are not eligible; patients who have a history of major depression that is controlled with chronic oral therapy are eligible provided they have no history of inpatient hospitalization, history of documented suicide attempt or ideations, and are managed with one anti-depressant which has not required dose adjustment in 6 weeks; patients with a history of depression who would otherwise be eligible should be evaluated by a mental health professional prior to enrollment if there is any uncertainty regarding the status of their mental health; Note: for patients with psychotropic treatments ongoing at baseline, the dose and the schedule should not be modified within the previous 6 weeks prior to start of study drug
* Patient has ≥ Common Terminology Criteria for Adverse Events (CTCAE) grade 3 anxiety
* Patient has other prior or concurrent malignancy (except for the following: adequately treated basal cell or squamous cell skin cancer, or other adequately treated in situ cancer, early gastric or GI cancer resected completely by endoscopy procedures or any other cancer from which the patient has been disease free for ≥ 3 years)
* Patient has a history of non-compliance to medical regimen or inability to grant consent
* Patient is concurrently using other approved or investigational antineoplastic agent
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test (> 5 milli-international unit [mIU]/mL); patients with elevated hCG at baseline that is judged to be related to the tumor are eligible if hCG levels do not show the expected doubling when repeated 5-7 days later, or pregnancy has been ruled out by vaginal ultrasound
* Patient who is not willing to apply highly effective contraception during the study and through the duration as defined below:

  * Sexually active males should use a condom during intercourse while taking drug and for 16 weeks after the final dose of study treatment and should not father a child in this period, but may be recommended to seek advice on conservation of sperm; a condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid
  * Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, must use highly effective contraception during the study and through at least 4 weeks after the final dose of study treatment
  * Highly effective contraception is defined as either:

    * Total abstinence: When this is in line with the preferred and usual lifestyle of the subject; (periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception)
    * Female sterilization: have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment; in case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male partner sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate); (for female study subjects, the vasectomized male partner should be the sole partner for that patient)
    * Use a combination of the following (both a+b):

      * a. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
      * b. Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository
      * c. Note: hormonal contraception methods (e.g. oral, injected, and implanted) are not allowed as buparlisib decreases the effectiveness of hormonal contraceptives
* Women are considered post-menopausal and not of child-bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) at least six weeks ago; for women with therapy-induced amenorrhea, oophorectomy or serial measurements of follicle stimulating hormone (FSH) and/or estradiol are needed to ensure postmenopausal status; Note: Ovarian radiation or treatment with a luteinizing hormone-releasing hormone (LH-RH) agonist (goserelin acetate or leuprolide acetate) is not permitted for induction of ovarian suppression
* Patients with a history of central nervous system involvement by CLL or who have prolymphocytic leukemia (PLL)
* Patients with known hepatitis B or hepatitis C (active or carriers)
* Patients with diarrhea ≥ CTCAE grade 2
* Patients who have received oral or IV chemotherapy or targeted anticancer therapy ≤ 2 weeks (4 weeks for nitrosourea, antibodies or mitomycin-C) prior to study enrollment; steroids used for anti-cancer properties must be tapered to 10 mg or less of prednisone (or equivalent) for at least 2 weeks prior to initiating therapy
* Patients who have received prior treatment with a pan-selective PI3K inhibitor are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-01; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of buparlisib when combined with ibrutinib in relapsed/refractory CLL for ibrutinib naive patients defined as the dose level at which no more than 1 of 6 patients experiences a dose-limiting toxicity | 28 days
  Adverse events and toxicities will be summarized using NCI CTCAE version 4 and based on severity and perceived attribution to study treatment.
MTD of buparlisib when combined with ofatumumab in relapsed/refractory CLL for ibrutinib pre-treated patients defined as the dose level at which no more than 1 of 6 patients experiences a dose-limiting toxicity | 28 days
  Adverse events and toxicities will be summarized using NCI CTCAE version 4 and based on severity and perceived attribution to study treatment.

SECONDARY OUTCOMES:
Complete response rate | Up to 5 years
  Reported descriptively in tabular form.
Incidence of non-dose limiting toxicities and adverse events | Up to 5 years
  Summarized by the NCI CTCAE version 4.03 criteria and tabulated across all patients who received any treatment with a focus on severe (grade 3+) adverse events and toxicities (those deemed at least possibly related to study treatment).
Nodal response rate | Up to 5 years
  Reported descriptively in tabular form.
Overall response rate | Up to 5 years
  Reported descriptively in tabular form.
Overall survival | Up to 5 years
  Calculated by the Kaplan-Meier method.
Progression-free survival | Up to 5 years
  Calculated by the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathon Cohen, MD, MS, Principal Investigator — Emory University
Locations (1):
- Emory University/Winship Cancer Institute, Atlanta, Georgia, United States